CLINICAL TRIAL: NCT00536445
Title: Use of Neurally Adjusted Ventilatory Assist (NAVA) in an Intubated Premature Infant: A Case Control Study on the Servoi Ventilator
Brief Title: Use of NAVA in Intubated Preterm
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Another institution performed the study
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr Michael Dunn, SHSC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 124-2007
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Infant, Premature; Respiration, Artificial
Keywords: NAVA; Preterm; Case study
MeSH Terms: conditions — Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NAVA — Neurally Adjusted Ventilatory Assist (mechanical ventilation controlled by the diaphragm electrical activity)
  Other Names: Servoi (Maquet Critical Care AB)

SUMMARY:
The present protocol will demonstrate the feasibility and efficacy of a newly developed mode of mechanical ventilation, Neurally Adjusted Ventilatory Assist, commonly known as NAVA. During NAVA, the timing and magnitude of pressure delivered are controlled by the infants' diaphragm electrical activity (EAdi), a validated measurement of neural respiratory drive. Recent clinical trials in adults and term infants have shown that NAVA is more synchronous than conventional pressure support ventilation, and that NAVA delivers lower mean airway pressures to achieve the same ventilation and respiratory muscle unloading. NAVA has recently been approved for use in neonates by Health Canada and the FDA in the United States, and is commercially available on the Servoi ventilator (Maquet Critical Care, Solna, Sweden). The present protocol is designed as a "case study" where the researchers responsible would like to evaluate the feasibility and efficacy of ventilating a premature baby on NAVA with the Servoi for 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborn (>1 day postnatal age, gestational age >23 weeks, birth weight <1250g), intubated and mechanically ventilated, and breathing spontaneously, as defined by the ability to trigger the ventilator. The infant should be breathing on conventional ventilation (SIMV, assist control, or pressure support) with the following ventilator parameters: assist control/pressure support < 22 cm H2O, PEEP 4-6 cm H2O Fi02<.30

Exclusion Criteria:

* Pneumothorax, degenerative neuromuscular disease, bleeding disorders, cardiovascular instability, cyanotic congenital cardiovascular disease, phrenic nerve damage/diaphragm paralysis, esophageal perforation, use of high frequency oscillatory or jet ventilation, contraindication to changing NG tube, or if infant is deemed "too unstable" by the clinical team. The use of narcotics is an exclusion criteria.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
• Patient-ventilator synchrony (trigger delays, cycling-off delays) • Phasic electrical activity of the diaphragm EAdi • Tonic EAdi • tidal volume, airway pressure, respiratory rate • Oxygen saturation, transcutaneous CO2, FIO2 | end of the 12 hour trial

SECONDARY OUTCOMES:
• Number of times back-up rate started (per hour) • Number of PEEP or NAVA level adjustments | end of the 12 hour trial

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunn, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Jennifer Beck, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- NICU, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Beck J, Campoccia F, Allo JC, Brander L, Brunet F, Slutsky AS, Sinderby C. Improved synchrony and respiratory unloading by neurally adjusted ventilatory assist (NAVA) in lung-injured rabbits. Pediatr Res. 2007 Mar;61(3):289-94. doi: 10.1203/01.pdr.0000257324.22406.93. PMID 17314685